CLINICAL TRIAL: NCT00650143
Title: Safety and Efficacy of Sitagliptin Plus Granulocyte-colony Stimulating Factor in Patients Suffering From Acute Myocardial Infarction
Brief Title: Sitagliptin Plus Granulocyte-colony Stimulating Factor in Acute Myocardial Infarction
Acronym: SITAGRAMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Hans Theiss, Professor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22021980
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Acute Myocardial Infarction
Keywords: Stem cell; Myocardial infarction; G-CSF; CD26-inhibition
MeSH Terms: conditions — Myocardial Infarction | interventions — Lenograstim; Sitagliptin Phosphate; Sodium Chloride; Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Application G-CSF (10µg/kg/d divided in two doses subcutaneously) over a period of 5 days and Sitagliptin 100 mg each day for 28 days.
  n=74
  Interventions: Drug: Lenograstim (GRANOCYTE)=GCSF; Drug: Sitagliptin (Januvia)
- 2 (Placebo Comparator): NaCl 0.9% applied twice daily over a period of 5 days and oral Placebo given once a day for 28 days.
  n=74
  Interventions: Drug: Sodium Chloride (NaCl) 0.9 %; Drug: Gelatin

INTERVENTIONS:
Drug: Lenograstim (GRANOCYTE)=GCSF — 10 µg/kg/d s.c. for 5 days divided in two dosages per day
  Arms: 1
Drug: Sitagliptin (Januvia) — 100 mg p.o. per day for 28 days
  Arms: 1
Drug: Sodium Chloride (NaCl) 0.9 % — applied s.c. twice a day for 5 days
  Arms: 2
Drug: Gelatin — One capsule p.o. per day for 28 days
  Arms: 2

SUMMARY:
Trial design:

This Phase III, investigator-driven, randomised, placebo-controlled efficacy and safety study will compare the effects of Sitagliptin in combination with granulocyte-colony stimulating factor (Lenograstim, G-CSF) on the improvement of myocardial function in patients undergoing routine percutaneous coronary revascularisation for acute myocardial infarction (time from onset of infarction to intervention 2 to 24 hours). The primary objective of this study is to compare between a treatment of G-CSF plus Sitagliptin, (G-CSF/Sitagliptin treatment group, n=87) versus Placebo (control treatment group, n=87) in change of global myocardial function from baseline to 6 months of follow-up.

DETAILED DESCRIPTION:
The trial will be conducted as a multi-centre trial. Secondary objectives of this study are to monitor changes of regional myocardial function, myocardial perfusion and extent of non-viable myocardium from baseline to 6 months after revascularisation between the treatment groups. Furthermore the following parameters over up to 12 months of follow-up are analysed: occurrence of major adverse cardiac events (death, myocardial infarction, coronary bypass grafting, or re-intervention), spontaneously reported adverse events. Analyses of cardiac function consists of evaluation of segmental systolic wall thickening, end-diastolic volume, end-systolic volume, stroke volume, ejection fraction and cardiac output by means of magnetic resonance imaging (MRI). The extent of non-viable myocardium and myocardial perfusion will be assessed using contrast enhanced MRI.

This study consists of a revascularisation period (angioplasty of the infarcted vessel), a treatment period (up to 28 days), and a follow-up period (up to 12 months). The Revascularisation Period starts with the treatment of the patient in the emergency room. As soon as possible the patient will be transferred to the catheterisation laboratory where acute percutaneous coronary intervention (PCI) of the infarct-related artery will be performed. The first phase of the Treatment Period consists of a screening period during which a patient's eligibility is preliminarily evaluated. The second phase of the Treatment Period is the randomisation for patients in the control or G-CSF/Sitagliptin treatment group. After baseline MRI, patients are randomised. Patients will be treated either with G-CSF (10µg/kg/d divided in two doses subcutaneously) over a period of 5 days and Sitagliptin 100 mg each day for 28 days or with placebo. Patients will be randomised in 1:1 ratio to the control and verum therapy treatment groups. Follow-up Period assessments will be performed in all patients at 6 months including clinical status, occurrence of adverse events, laboratory investigations, and MRI. To assess occurrence of in-stent restenosis, routine control angiography will be performed in all patients 6 months after initial PCI. Safety will be evaluated by monitoring treatment-emergent signs and symptoms, 12-lead ECGs, vital signs, physical examination, and clinical laboratory assessments after 1 month and 1 year.

ELIGIBILITY:
Inclusion criteria

1. Be at least 18 years old, male or female
2. Have acute ST segment elevation myocardial infarction (typical chest pain of more than 30 minutes duration, presence of ST-segment elevation in at least two contiguous leads or left bundle-branch block) and/or occluded coronary artery
3. Intervention of infarct related artery by PCI/Stenting within 2-24 hours after onset of acute myocardial infarction.
4. have creatinin kinase elevation of more than three times of upper normal level (i.e. 540 U/l) accompanied by a significant elevation of CK-MB isoenzyme and/or Troponin I/T
5. Have regional wall motion abnormality (comprising hypo-, a- or dyskinesia) of at least one myocardial segment demonstrated with MRI.
6. Patients who are further suitable for coronary angiography and angioplasty with stenting of the infarct related artery.
7. Have the ability to understand the requirements of the study, and agree and be able to return for the required assessments.
8. Give a written informed consent.

Exclusion criteria

General:

1. Women of childbearing potential, pregnancy or being lactating.
2. Be unable to undergo percutaneous cardiac catheterisation
3. Have contraindications against magnetic resonance imaging (e.g. non-MR compatible implants or medical devices)
4. Have conditions that may severely degrade image quality (e.g. severe arrhythmia) or prevents from MR scanning (e.g. claustrophobia)
5. Previous enrolment in the present trial or administration of any study medication within the previous 30 days. Study drug is defined as any material (placebo or drug) dispensed under the provisions of a protocol.
6. Have other severe concurrent illness (e.g., active infection, malignancy).
7. Life expectancy of less than one year.
8. Have a history of alcohol or drug abuse within 3 months prior to admission or factors jeopardising follow-up.

Renal, hepatic, metabolic:

1. Moderate to severe renal impairment (Crea level >1.7 mg/dL or glomerular filtration rate <35 ml/min).
2. Diabetes type 1 patients.
3. Diabetic ketoacidosis.
4. Concomitant medications known to cause hypoglycemia, such as sulfonylureas.
5. Severe liver dysfunction.

Haematologic:

1. Malignant haematological diseases, i.e. chronic myeloic leukemia (CML) or myelodysplastic syndromes (MDS)
2. Severe congenital neutropenia with cytogenetic abnormalities
3. Known allergic reaction vs. Lenograstim

Cardiovascular:

1. Acute cardiogenic shock
2. Cardiomyopathy with an ejection fraction below 0.25 (i.e. ischemic or dilated cardiomyopathy resulting in congestive heart failure)
3. Infective endocarditis
4. Factors contraindicating cardiac catheterisation (e.g. severe allergy against iodine, severe thyroid disease)
5. Planned operative revascularisation
6. Left ventricular thrombus
7. Severe cardiac arrhythmias (i.e. malignant sustained or non-sustained ventricular tachycardia or ventricular fibrillation) within 24 hours after admission.

Pulmonary:

1. Acute massive pulmonary infiltrations
2. History of pneumonia in the last 4 weeks

Other:

1. Therapy with immunosuppressants, cytostatics, corticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change of global myocardial function from baseline to 6 months of follow-up. | Recruitment period: 4,5 years. Follow-up assessment: 1 year. Analyses and reporting: 6 months. Overall duration: 6 years.

SECONDARY OUTCOMES:
Segmental end-diastolic myocardial thickness, segmental systolic wall thickening, regional contractile reserve, end-diastolic and end-systolic volumes, stroke volume, and cardiac output in MRI | 6 months of follow-up
Extent of non-viable myocardium will be monitored from baseline up to 6 months measured by MRI delayed enhancement. | 6 months follow up
Change of myocardial perfusion at rest up to 6 months as measured by signal-time curve parameters using first-pass perfusion MRI | 6 month follow up
Occurrence of major adverse cardiac events (death, myocardial infarction, CABG, or re-intervention) up to 12 months. | 12 months follow up
Safety of a treatment of Sitagliptin in combination with G-CSF in CAD patients suffering from MI (spontaneously reported adverse events (AEs) up to 12 months). | 12 months follow up
Change of peripheral blood stem cell populations: CD34, CD34/KDR and CD34/CD26 positive cells prior to and 5 days after therapy initiation. | 1 week follow up
Change of plasma levels of NT-pro-BNP, glucose, complete blood count, CRP, platelets, CK, cTnI prior to and 5 and 28 days, and 6 months after therapy initiation | 12 month follow up
Assessment of in stent restenosis using angiography 6 months after facultative PCI | 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang M Franz, Prof. Dr., Principal Investigator — Clinic of the University of Munich-Grosshadern, Department of Cardiology
Locations (1):
- Clinic of the University of Munich-Grosshadern, Department of Cardiology, Munich, Germany

REFERENCES:
- [Background] Engelmann MG, Theiss HD, Hennig-Theiss C, Huber A, Wintersperger BJ, Werle-Ruedinger AE, Schoenberg SO, Steinbeck G, Franz WM. Autologous bone marrow stem cell mobilization induced by granulocyte colony-stimulating factor after subacute ST-segment elevation myocardial infarction undergoing late revascularization: final results from the G-CSF-STEMI (Granulocyte Colony-Stimulating Factor ST-Segment Elevation Myocardial Infarction) trial. J Am Coll Cardiol. 2006 Oct 17;48(8):1712-21. doi: 10.1016/j.jacc.2006.07.044. Epub 2006 Sep 11. PMID 17045910
- [Derived] Brenner C, Adrion C, Grabmaier U, Theisen D, von Ziegler F, Leber A, Becker A, Sohn HY, Hoffmann E, Mansmann U, Steinbeck G, Franz WM, Theiss HD. Sitagliptin plus granulocyte colony-stimulating factor in patients suffering from acute myocardial infarction: A double-blind, randomized placebo-controlled trial of efficacy and safety (SITAGRAMI trial). Int J Cardiol. 2016 Feb 15;205:23-30. doi: 10.1016/j.ijcard.2015.11.180. Epub 2015 Nov 30. PMID 26709136